CLINICAL TRIAL: NCT02318641
Title: Measurement of the Oxygen Saturation in the Retinal Vessels With Oxymap
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kagawa University (Other)
Responsible Party: Principal Investigator, Akitaka Tsujikawa, Professor and Chairman, Kagawa University
Other Study IDs: H26-046
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Chorioretinal Disorders in Diseases Classified Elsewhere
Keywords: oxygen consumption; retinal oximetry
MeSH Terms: interventions — Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: oximetry — Retinal oximetry will be performed with Oxymap.

SUMMARY:
Retinal oximetry can be measured with newly developed Oxymap (Oxymap ehf, Reykjavik, Iceland). Briefly, the device simultaneously acquires digital images at two wavelengths and automatically tracks retinal vessels on both images. Retinal vessel oxygen saturation is estimated by spectrophotometric analysis of light reflected from retinal vessels and from the immediately surrounding retina. Oxygen saturation measurements are made on major temporal arteries and veins. Briefly, the first and second degree vessels are used, with the addition of third degree vessels in images where peripapillary haemorrhage prevented analysis close to the optic disc. Vessel segments chosen for analysis are used consistently for consecutive measurements in the same retina.

DETAILED DESCRIPTION:
Retinal oximetry can be measured with newly developed Oxymap (Oxymap ehf, Reykjavik, Iceland). Briefly, the device simultaneously acquires digital images at two wavelengths and automatically tracks retinal vessels on both images. Retinal vessel oxygen saturation is estimated by spectrophotometric analysis of light reflected from retinal vessels and from the immediately surrounding retina. Oxygen saturation measurements are made on major temporal arteries and veins. Briefly, the first and second degree vessels are used, with the addition of third degree vessels in images where peripapillary haemorrhage prevented analysis close to the optic disc. Vessel segments chosen for analysis are used consistently for consecutive measurements in the same retina.

Retinal oximetry in various chorioretinal diseases will be measured with Oxymap.

ELIGIBILITY:
Inclusion Criteria:

* Healthy eyes and eyes with various chorioretinal diseases, including diabetic retinopathy, retinal vein occlusion, epiretinal membrane, macular hole, inherited chorioretinal diseases, glaucoma, retinal detachment, etc.

Exclusion Criteria:

* Eye with medial opacity.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy eyes and eyes with various chorioretinal disease.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change of retinal oxygen saturation from baseline at 6 months | Six months.

CONTACTS AND LOCATIONS:
Overall Officials: AKITAKA TSUJIKAWA, MD, Principal Investigator — Kagawa Univerisity Faculty of Medicine
Locations (1):
- Kagawa University Faculty of Medicine, Hiragi, Kagawa-ken, Japan